CLINICAL TRIAL: NCT00984854
Title: A Trial to Investigate the Clinical Safety, Local Toleration, and Systemic Pharmacokinetics of Repeated, Escalating Concentrations of Intradermal RN1004 to Wounds of Healthy Subjects.
Brief Title: Investigation Into the Safety of Intradermal Juvidex (M6P) Administered to Wounds of Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: John Hutchison, Medical Director, Renovo
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RN1004-319-1001
Record Dates: First submitted 2009-09-24; First posted 2009-09-25 (Estimated); Last update posted 2009-09-25 (Estimated); Status verified 2009-09

CONDITIONS: Cicatrix; Re-epithelialisation
Keywords: Cicatrix; Scar; Wound-healing; Re-epithelialisation; RN1004; Mannose-6-phosphate; M6P; Juvidex
MeSH Terms: conditions — Cicatrix | interventions — mannose-6-phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intradermal Juvidex (Experimental)
  Interventions: Drug: Juvidex
- Placebo (vehicle) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Juvidex — Intradermal Juvidex, 100μl of 50mM (1.41mg/100μl) administered just prior to wounding and 200μl administered 24 h later
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 100mM (2.82mg/100μl) administered just prior to wounding and 200μl administered 24 h later
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 200mM (5.64mg/100μl) administered just prior to wounding and 200μl administered 24 h later
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 300mM (8.46mg/100μl) administered just prior to wounding and 200μl administered 24 h later
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 400mM (11.28mg/100μl) administered just prior to wounding and 200μl administered 24 h later
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Juvidex — Intradermal Juvidex, 100μl of 600mM (16.93mg/100μl) administered just prior to wounding and 200μl administered 24 h later
  Other Names: Mannose-6-phosphate; M6P; RN1004
  Arms: Intradermal Juvidex
Drug: Placebo — Intradermal Placebo (0.9% phosphate buffered saline, pH 7.0), 100μl administered just prior to wounding and 200μl administered 24 later
  Arms: Placebo (vehicle)

SUMMARY:
The purpose of this study was to investigate the safety and toleration of various doses of intradermal Juvidex (mannose-6-phosphate) administered to punch biopsies of normal subjects.

DETAILED DESCRIPTION:
Each subject received a total of four wounds, two 3mm punch biopsies (at least 5cm apart) to the upper, inner aspect of each arm.

Subjects served as their own control, i.e. one punch biopsy on Arm 1 received Juvidex and the other punch biopsy received Placebo or Standard Care. Arm 2 punch biopsies received the same treatments as for Arm 1 but in reverse, i.e. treatments were matched across the arms.

On Day 0 the two areas for punch biopsies on Arm 1 were marked and anaesthetised and randomised to receive Juvidex or Placebo. Prior to wounding sites were injected intradermally with 100μl investigational product per site. Juvidex was dosed at 50, 100, 200, 300, 400, and 600mM.

On Day 1 (24 h later) wounds were dosed as on Day 0 but with 200μl investigational product per site. On Day 3 the biopsy sites on Arm 1 were excised to determine re-epithelialisation.

Arm 2 treatments and punch biopsies were carried out on Day 3, with further dosing 24 h later on Day 4 (as with Arm 1 wounding and treatments). These biopsy sites were excised on Day 8 of the study to obtain a 5 day-old wound.

The randomisation of the treatment allowed for control of possible positional effects on healing. One subject in each group was randomised to receive only Placebo and Standard Care to their biopsy wounds.

ELIGIBILITY:
Inclusion Criteria:

* Clinically healthy male and female subjects aged 18-45 years inclusive
* Weight between 40 and 150kg and a BMI within the permitted range for their height using Quetelet's index - weight (kg)/height²(m). The permitted index is between 15 - 55 kg/m2

Exclusion Criteria:

* Subjects who on direct questioning and physical examination have history or evidence of hypertrophic or keloid scarring or with tattoos or previous scars in the area to be biopsied
* Subjects who have had surgery in the area to be biopsied within the previous 12 months
* Afro-Caribbean subjects are excluded because of the increased susceptibility to hypertrophic and keloid scarring
* Subjects, who on direct questioning and physical examination, have evidence of any past or present clinically significant disease, particularly coagulation disorders, diabetes, immuno-mediated conditions and skin diseases and allergies, such as clinically significant eczema
* Subjects with a history of clinically significant allergies, especially drug hypersensitivity to lignocaine or allergy to surgical dressings to be used in this trial; or to any excipients or vehicle in the formulation or delivery vehicle
* Subjects with any clinically significant abnormality following review of pre-trial laboratory data and physical examination
* Subjects who are taking, or have taken, certain prescribed drugs in the four weeks prior to Day 0 and in particular topical or systemic steroids, anti-inflammatory, anti-coagulant, antiproliferative drugs and antibiotics Certain drugs are not excluded in this trial, including OTC analgesics such as paracetamol and codeine, vitamin and mineral supplements and OTC cold remedies and hormonal contraceptives. If antibiotics are required after Day 0, this will not exclude subjects from continuation in this trial and the data will be recorded in the CRF
* Subjects who have taken part in a clinical trial within 3 months prior to admission to this trial, or who are currently participating in a clinical trial, whether an investigational drug was involved or not
* Subjects who have any clinical evidence of severe ongoing or prolonged depression or mental illness
* Subjects who smoke more than 20 cigarettes a day
* Subjects who drink more than 28 units of alcohol per week (1 unit = 1/2 pint of beer (285mls) or 25ml of spirits or 1 glass of wine)
* Subjects who have evidence of drug abuse
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B surface antigen or hepatitis C antibody. Subjects with previous vaccination against Hepatitis B are not excluded per se
* Subjects who are known to have or had serum hepatitis or who are carriers of the hepatitis B core antibody and who show less than 10 units per litre of Anti-HBs, (unless deemed NOT to be a hepatitis B carrier by the local Public Health laboratory)
* Subjects who have previously had a positive result to the test for HIV antibodies, or who admit to belonging to a high-risk group
* Subjects who are pregnant or planning to get pregnant or lactating or not taking adequate contraceptive precautions. Subjects must use suitable mechanical forms of contraception (or abstinence) during the trial
* Subjects who are receiving the following drugs: cyclosporine, cyclophosphamide, taxol or warfarin
* Subjects who have pre-existing clinically significant neurological conditions
* In the opinion of the Investigator, a subject who is not likely to complete the trial for whatever reason

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2004-01; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
To assess the safety and local toleration of various dose levels of Juvidex (RN1004) injected intradermally in healthy volunteers. | 22 Days

SECONDARY OUTCOMES:
To determine the systemic PK of various dose levels of Juvidex injected intradermally. | 22 days
To determine the histological effects on wound healing (re-epithelialisation, inflammatory cell infiltrate, angiogenesis and matrix deposition) of intradermal injections of Juvidex in healthy subjects. | Day 3 and 5
To find the maximum tolerated dose (MTD) of Juvidex | 22 days

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Bond, Principal Investigator — Renovo; Jonathan Duncan, Principal Investigator — Renovo
Locations (1):
- Renovo, Manchester, United Kingdom